CLINICAL TRIAL: NCT06843252
Title: Home-based TDCS for Cognitive and Behavioral Symptoms in Huntington's Disease: a Pilot Feasibility and Mechanistic Study
Brief Title: Home-based TDCS (Transcranial Direct Current Stimulation) for Cognitive and Behavioral Symptoms in Huntington's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Huntington's Disease Society of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: STUDY00000882
Record Dates: First submitted 2025-01-24; First posted 2025-02-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Huntington Disease
Keywords: Transcranial direct current stimulation; Home-based; Behavioral symptoms; Cognitive symptoms
MeSH Terms: conditions — Huntington Disease; Behavioral Symptoms; Neurobehavioral Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blind cross-over clinical trial. Participants will be their own control and in addition, caregivers will provide collateral information regarding the participant via structured interviews or questionnaires.
Who Masked: Participant, Investigator
Masking Description: Patients will be blinded throughout the trial. As the application of tDCS electrical current over the skin can be perceived by the participants, the study team will employ a sham condition that has been shown to be reliable and indistinguishable from active treatment in previous clinical trials published in the available scientific literature. An individual on the study team will be delegated to randomize and program and re-program devices. Participants will act as their own control. The researcher supervising the stimulation will be blinded to the intervention the participant is receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active TDCS treatment (Experimental): The active-tDCS treatment will consist of a constant 2mA current applied during 30-minute sessions with a 30 second ramp up and ramp down at the start and end of the stimulation.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham TDCS treatment (Sham Comparator): Sham-tDCS treatment will consist of the same montage as the active TDCS with the built-in function of the device that has been shown to be indistinguishable from the active treatment in previous trials described in the literature.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — The active-tDCS treatment will consist of a constant 2mA current applied during daily 30-minute sessions with a 30 second ramp up and ramp down at the start and end of the stimulation. The anode electrode will be placed over the left dorsolateral prefrontal cortex (DLPFC) and the cathode electrode over the right DLPFC.
  Other Names: tDCS
  Arms: Active TDCS treatment
Device: Sham tDCS — Sham-tDCS treatment will consist of the same montage as the active TDCS with the built-in function of the device that has been shown to be indistinguishable from the active treatment in previous trials described in the literature.
  Other Names: Control
  Arms: Sham TDCS treatment

SUMMARY:
The researchers hope to find out effects of transcranial direct current stimulation (tDCS) sessions on the behavioral symptoms of Huntington's Disease. If participants are eligible to continue, they will be provided a device to administer the tDCS for 30 minutes each day and be asked to answer questions with the study staff . Participants will be asked to return to the study center for follow ups and to undergo additional cognitive tests and questionnaires. Participants will also be asked to answer questionnaires via a web conferencing platform (Zoom) during the course of the study. Caregivers of the participants will be asked to answer questionnaires to collect more information about the participants.

DETAILED DESCRIPTION:
This clinical trial will investigate the effects of transcranial direct current stimulation (tDCS) over cognitive and behavioral symptoms of patients with Huntington's disease (HD). The study will also investigate underlying neurobiological mechanisms of tDCS in HD.

ELIGIBILITY:
Inclusion Criteria:

1. individuals aged 18-85 years with confirmed HD mutation and/or established family history alongside typical symptoms (i.e., chorea) of HD;
2. early (stages 1 and 2) or moderate (stage 3) stages according to Shoulson-Fahn criteria, also known as the UHDRS total functional capacity (TFC) scale (Bates, Tabrizi, and Jones 2014);
3. exhibit mild to moderate behavioral symptoms defined by severity scores in the PBA-S between 1 and 3 for any of the evaluated symptoms and no symptoms with a severity score of 4;
4. stable doses of medications for at least one month.
5. Ability of subject to understand and the willingness to sign a written informed consent document.
6. Have a caregiver willing to be present during tDCS sessions and answer questionnaires.

Caregiver

1. An adult who serves as an unpaid caregiver for an individual enrolled in the study as interpreted by the PI or delegate physician.
2. Adequate cognitive capacity to provide verbal consent to participate in the caregiver arm of the study.
3. Adequate reading, writing, hearing, and verbal capacity to provide collateral information about the study participant as well as answer questions related to their health and care.

Exclusion Criteria:

1. Unstable medical conditions (e.g. unstable angina, uncontrolled diabetes and hypertension, advanced cancer, etc.);
2. History of epilepsy;
3. Clinical diagnosis of major cognitive disorder (i.e., dementia);
4. Have risk of suicidal behavior, defined as any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the 3 months prior to screening (Posner et al. 2011);
5. Being an active participant in other therapeutic clinical trial;
6. Determined to be incapable of consent per PMH or via assessment by the study staff at time of consent.
7. Participant has a pacemaker or any other implanted device/material contraindicated in the use of tDCS per current labeling requirements.

Caregiver

1. Any individual who does not meet all the inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants that met Inclusion Criteria | Baseline
  Percentage of participants screened that met Inclusion Criteria
Percentage of Participants that Agreed to Randomization | Baseline
  Percentage of eligible participants that were screened and met eligibility that agreed to be randomized.
Completed period 1 of study | Day 13
  Percentage of participants who completed first 2 weeks of treatment or sham
Completed period 2 of study | Day 35
  Percentage of participants that completed both the first period, the washout period and the second period of the study
Completion of study to last visit | Day 36 (or day 37)
  Percentage of participants that completed study from randomization to tDCS/Sham crossed over to alternate treatment/sham and returned for final visit
TDCS Acceptability Scale | Day 14 and Day 35
  This Likert scale scores 10 items for user acceptability. Each item is scored from 0-10 giving. Some items have negative valence, in which lower scores indicate higher acceptability. An averaged of adjusted scores for all items is calculated to produce a global acceptability score ranging from 0 to 10. A higher score on the global score indicates better acceptability.
tDCS Side Effects Scale | Day 8, 14, 29 and 35
  This Likert scale includes 10 items scored from 0-10 for possible side effects. The first 9 items include a list of possible side effects and the last item is free field for the report of any additional side effects. Lower scores indicate less intensity of side effects. Scores will be reported for each individual item.

SECONDARY OUTCOMES:
Problem Behaviors Assessment Scale (PBA-S) | Baseline, and days 14, 22, and 35.
  This scale rates the participant's average behavior over the past weeks by taking into account the severity and frequency of a range of psychiatric symptoms. There are 11 items assessed with a possible total score range of 0-176. A lower score indicates less psychiatric symptoms.
Frontal Assessment Battery (FAB) | Baseline, and days 14 and 35.
  This scale is a brief cognitive and behavioral battery. The total maximum score is 18, with higher scores indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Macedo e Cordeiro, MD, MSc, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at the Glenn Bigs Institute for Alzheimer's and Neurodegenerative diseases at UT Health San Antonio. After the study is completed, the de-identified, archived data will be transmitted to and stored at the Glenn Bigs Institute for Alzheimer's and Neurodegenerative diseases at UT Health San Antonio, for use by other researchers including those outside of the study. Permission to transmit data to the Glenn Biggs Institute for Alzheimer's and Neurodegenerative diseases at UT Health San Antonio will be included in the informed consent.
Supporting Information: Study Protocol, SAP
Time Frame: When the study is completed and data is analyzed.